CLINICAL TRIAL: NCT00340288
Title: Fibroid Growth Study
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901209; 01-E-N209
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Uterine Leiomyomas
Keywords: Neoplasms; Life Style/Endrocrinology; Magnetic Resonance Imaging; Molecular Characterization; Leiomyoma
MeSH Terms: conditions — Myofibroma; Neoplasms; Leiomyoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Premenopausal fibroid cases: Premenopausal women (18 years or older) with at least one uterine leiomyoma diagnosis confirmed by ultrasound

SUMMARY:
Uterine leiomyomas, commonly called fibroids, are a major health concern for women of reproductive age. The objectives of the study described herein are to investigate the growth dynamics of uterine leiomyomas in a clinically relevant population of women. We will test the hypotheses that uterine leiomyomas are heterogeneous in terms of their growth characteristics and in their clinical symptoms or outcomes, and that differences in leiomyoma growth dynamics can be discriminated by molecular markers and cellular phenotypes. Participants will include 300 premenopausal women (greater than 18 years old) with at least one uterine leiomyoma. The inclusion criteria for patient enrollment is confirmed diagnosis of leiomyoma by ultrasound. At least one leiomyoma must be equal to or greater than 2 cm in diameter and the uterus must be enlarged to the size typical during the eigth week of pregnancy. After enrollment and informed consent, T1- and T2-weighted magnetic resonance image (MRI) scans will be conducted beginning at the first visit and then at 3, 6, and 12 months. Each patient will have a physical exam, provide urine and blood samples at each MRI visit, and respond to an initial extensive telephone-administered questionnaire followed by abbreviated monthly questionnaire updates. A number of the enrolled women will require surgical intervention (hysterectomy/myomectomy) as standard care. If surgery is an outcome for women enrolled in the study, MRI will be conducted before surgery and the surgical pathologist will map uterine leiomyomas for comparison to MRI. Leiomyoma samples will be analyzed for histopathological and molecular changes correlated with growth. Because hysterectomy and myomectomy are common outcomes in women with leiomyomas, we anticipate tissue will be available from at least 100 of the 300 women in the study. For those women who opt for surgery, we will also administer a brief (less than 5 minute) questionnaire clarifying their reason for electing surgery. Upon completion of data collection, we will be able to compare leiomyoma growth as a function of multiplicity and location; examine the relationship between leiomyoma growth and clinical symptoms or outcome; identify molecular, cellular, and pathological characteristics of leiomyomas with differing growth dynamics; and examine endocrinological parameters and lifestyle factors related to differential growth dynamics of uterine leiomyomas. The data may be used to establish a clinical severity scale and establish diagnostic markers currently not available for uterine leiomyomas.

DETAILED DESCRIPTION:
Uterine leiomyomas, commonly called fibroids, are a major health concern for women of reproductive age. The objectives of the study described herein are to investigate the growth dynamics of uterine leiomyomas in a clinically relevant population of women. We will test the hypotheses that uterine leiomyomas are heterogeneous in terms of their growth characteristics and in their clinical symptoms or outcomes, and that differences in leiomyoma growth dynamics can be discriminated by molecular markers and cellular phenotypes. Participants will include 300 premenopausal women (greater than 18 years old) with at least one uterine leiomyoma. The inclusion criteria for patient enrollment is confirmed diagnosis of leiomyoma by ultrasound. At least one leiomyoma must be equal to or greater than 2 cm in diameter and the uterus must be enlarged to the size typical during the eigth week of pregnancy. After enrollment and informed consent, T1- and T2-weighted magnetic resonance image (MRI) scans will be conducted beginning at the first visit and then at 3, 6, and 12 months. Each patient will have a physical exam, provide urine and blood samples at each MRI visit, and respond to an initial extensive telephone-administered questionnaire followed by abbreviated monthly questionnaire updates. A number of the enrolled women will require surgical intervention (hysterectomy/myomectomy) as standard care. If surgery is an outcome for women enrolled in the study, MRI will be conducted before surgery and the surgical pathologist will map uterine leiomyomas for comparison to MRI. Leiomyoma samples will be analyzed for histopathological and molecular changes correlated with growth. Because hysterectomy and myomectomy are common outcomes in women with leiomyomas, we anticipate tissue will be available from at least 100 of the 300 women in the study. For those women who opt for surgery, we will also administer a brief (less than 5 minute) questionnaire clarifying their reason for electing surgery. Upon completion of data collection, we will be able to compare leiomyoma growth as a function of multiplicity and location; examine the relationship between leiomyoma growth and clinical symptoms or outcome; identify molecular, cellular, and pathological characteristics of leiomyomas with differing growth dynamics; and examine endocrinological parameters and lifestyle factors related to differential growth dynamics of uterine leiomyomas. The data may be used to establish a clinical severity scale and establish diagnostic markers currently not available for uterine leiomyomas.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women included in the study must be at least 18 years if age, premenopausal, speak English, and have one or more uterine leiomyomas at least 2 cm in diameter and the utuerus must be enlarged to the size typical during the 8th week of pregnancy. Note that while the selcetion criteia are set to recruit women in which surgical intervention is a likely outcome, surgery is not a requirement for study inclusion.

EXCLUSION CRITERIA:

Women will be excluded if they are pregnant because of potential safety concerns associated with imaging and image contrast enhancements. If women become pregnant during the study, they wil have the option to stay in the study, but will have pelvic ultrasound scans in place of MRI scans.

Women who are taking or likely to start taking GnRH therapy will be excluded because this therapy, which is used as a treatment method for leiomyomas, sometmes induces their regression.

Women who are greater than 52 inches in circumference or greater than 350 pounds will be excluded because they will be too large to fit in the imaging equipment.

Women that have an intra-uterine device (IUD) will be excluded because these metal devices create 'shadowing' in MR images, making accurate measurement and interpretation of leiomyomas in the MRIs difficult.

Women are not excluded if they had a prior myomectomy, or if they are taking oral contraceptives.

The inclusion of only women of premenopausal age (greater than 18 years old) in this study is dictated by the nature of the condition.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Premenopausal women (18 years or older) with at least one uterine leiomyoma diagnosis confirmed by ultrasound. At least one fibroid must be equal to or greater than 2 cm in diameter and the uterus must be enlarged to the size typical during the eighth week of pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2001-06-27; Primary Completion 2006-04-01 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Size of fibroids as seen in MRI scans | 0, 3, 6, and 12 months after enrollment (1 year or through time of myomectomy or hysterectomy surgery)
  leiomyoma growth dynamics

SECONDARY OUTCOMES:
Symptomatology - bleeding and pain | 0, 3, 6, and 12 months after enrollment (1 year or through time of myomectomy or hysterectomy surgery)
  leiomyoma growth dynamics

CONTACTS AND LOCATIONS:
Overall Officials: Donna D Baird, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- University of North Carolina Medical Center, Chapel Hill, North Carolina, United States